CLINICAL TRIAL: NCT00238875
Title: A Phase II Study of Stereotactic Body Radiation Therapy in Patients With T1N0M0 Non-small Cell Lung Cancer (JCOG0403)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0403; C000000029
Record Dates: First submitted 2005-10-13; First posted 2005-10-14 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: T1N0M0 Non-small Cell Lung Cancer
Keywords: stereotactic body radiation therapy; T1N0M0 non-small cell lung cancer; radiotherapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Procedure/Surgery: stereotactic body radiation therapy
  Interventions: Procedure: stereotactic body radiation therapy

INTERVENTIONS:
Procedure: stereotactic body radiation therapy — Procedure/Surgery: stereotactic body radiation therapy

SUMMARY:
To evaluate the efficacy and safety of SBRT for T1N0M0 non-small cell lung cancer

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of SBRT for T1N0M0 non-small cell lung cancer，the following questions should be answered. Can SRT be an alternative standard treatment modality for inoperable patients? Can SRT can be a comparable standard treatment modality with lobectomy for operable patients? 12 Gy is the daily dose at the isocenter，and 48 Gy in total by 4 fractions will be irradiated by stereotactic irradiation over 4 to 8 days.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or transbronchoscopic cytologically confirmed non-small cell lung cancer
2. Stage IA with images within 28 days
3. No other intrathoracic lesions
4. Dose constraints of the organs at risk seem to be limited within range
5. Operable (Standard or Limited surgery) or Inoperable
6. Age>=20
7. No previous thoracic radiation
8. No previous chemotherapy
9. ECOG PS=0-2
10. Respiratory function (<=14 days) PaO2>=60 torr FEV1.0>=700 ml
11. Written informed consent

Exclusion Criteria:

1. No apparent radiation pneumonitis and fibrosis
2. No active tuberculosis without oral drugs
3. No double cancer
4. No pregnancy
5. No psychiatric disorder
6. No steroid administration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2004-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
3-years overall survival | During the study conduct

SECONDARY OUTCOMES:
Overall survival | During the study conduct
relapse-free survival | During the study conduct
local-relapse free survival | During the study conduct
3-years local relapse free survival | During the study conduct
patterns of relapse | During the study conduct
acute complications | within 8 weeks from starting treatment day
late complications | after 8 weeks from starting treatment day
serious complication rate | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Hiraoka, MD, PhD, Study Chair — Kyoto Universlty Hospital
Locations (16):
- Japan (16):
  - Kyushu University Hospital, Fukuoka,Higashi-ku,Maidashi,3-1-1, Fukuoka
  - Hiroshima University, School of Medicine, Hiroshima,Minami-ku,Kasumi,1-2-3, Hiroshima
  - Hokkaido University Hospital, North-14 West-5 Kita-ku,Sapporo, Hokkaido
  - Sapporo Medical University, S-1,W-16,Chuo-ku,Sapporo, Hokkaido
  - Institute of Biomedical Research and Innovation Hospital, Kobe,Chuo-ku,Minatojima-Minamimachi,2-2, Hyōgo
  - Kitasato University School of Medicine, Sagamihara,Kitasato,1-15-1, Kanagawa
  - Kyoto Universlty Hospital, Kyoto,Sakyoku,Shogoin,Kawahara-cho,54, Kyoto
  - Tohoku University Hospital, Sendai,Aoba-ku,Seiryo-machi,1-1, Miyagi
  - Tenri Hospital, Tenri,Mishima-cho,200, Nara
  - The University of Tokyo Hospital, Bunkyo-ku,Hongo,7-3-1, Tokyo
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-ku,Honkomagome,3-18-22, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku,Oyaguchikamimachi,30-1, Tokyo
  - Cancer Institute Hospital, Koto-ku,Ariake,3-10-6, Tokyo
  - Tokyo Women's Medical University, Shinjuku-ku,Kawada-cho,8-1, Tokyo
  - Keio University Hospital, Shinjuku-ku,Shinanomachi,35, Tokyo
  - University of Yamanashi Faculty of Medicine, Nakakoma,Tamaho,Shimokato,1110, Yamanashi

REFERENCES:
- [Background] Nagata Y, Negoro Y, Aoki T, Mizowaki T, Takayama K, Kokubo M, Araki N, Mitsumori M, Sasai K, Shibamoto Y, Koga S, Yano S, Hiraoka M. Clinical outcomes of 3D conformal hypofractionated single high-dose radiotherapy for one or two lung tumors using a stereotactic body frame. Int J Radiat Oncol Biol Phys. 2002 Mar 15;52(4):1041-6. doi: 10.1016/s0360-3016(01)02731-6. PMID 11958900
- [Background] Nagata Y, Takayama K, Matsuo Y, Norihisa Y, Mizowaki T, Sakamoto T, Sakamoto M, Mitsumori M, Shibuya K, Araki N, Yano S, Hiraoka M. Clinical outcomes of a phase I/II study of 48 Gy of stereotactic body radiotherapy in 4 fractions for primary lung cancer using a stereotactic body frame. Int J Radiat Oncol Biol Phys. 2005 Dec 1;63(5):1427-31. doi: 10.1016/j.ijrobp.2005.05.034. Epub 2005 Sep 19. PMID 16169670
- [Derived] Nagata Y, Hiraoka M, Shibata T, Onishi H, Kokubo M, Karasawa K, Shioyama Y, Onimaru R, Kozuka T, Kunieda E, Saito T, Nakagawa K, Hareyama M, Takai Y, Hayakawa K, Mitsuhashi N, Ishikura S. Prospective Trial of Stereotactic Body Radiation Therapy for Both Operable and Inoperable T1N0M0 Non-Small Cell Lung Cancer: Japan Clinical Oncology Group Study JCOG0403. Int J Radiat Oncol Biol Phys. 2015 Dec 1;93(5):989-96. doi: 10.1016/j.ijrobp.2015.07.2278. Epub 2015 Nov 11. PMID 26581137
- See also: Related Info — http://www.jcog.jp/